CLINICAL TRIAL: NCT06024161
Title: Weight Change and the Risk of Chronic Pain Following Hip and Knee Arthroplasties: A Nationwide Registry-based Cohort Survey Study.
Brief Title: Weight Change and the Risk of Chronic Pain Following Hip and Knee Arthroplasties
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Saber Muthanna Saber, MD, PhD fellow, Bispebjerg Hospital
Other Study IDs: p-2023-14578
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Persistent Postsurgical Pain; Arthritis Knee; Arthropathy of Knee; Arthropathy of Hip; Weight Loss; Weight Gain; Obesity
MeSH Terms: conditions — Pain, Postoperative; Weight Loss; Weight Gain; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Weight gainers: Weight gain 11-15 months after arthroplasty
  Interventions: Other: Weight gain
- Weight losers: Weight loss11-15 months after arthroplasty
  Interventions: Other: Weight loss
- Weight unchanged: Weight unchanged 11-15 months after arthroplasty
  Interventions: Other: Weight unchanged

INTERVENTIONS:
Other: Weight gain — ≥5% weight gain
  Groups: Weight gainers
Other: Weight loss — ≥5% weight loss after arthroplasty
  Groups: Weight losers
Other: Weight unchanged — <5% weight change after arthroplasty
  Groups: Weight unchanged

SUMMARY:
The study is a nationwide, register-based cohort survey study. The objective of this study is to investigate whether weight change is associated with the incidence of persistent postoperative pain following total hip arthroplasty and knee arthroplasty across non-obese and obese and patients.

ELIGIBILITY:
Inclusion Criteria:

- Patients operated with primary hip or knee arthroplasty for osteoarthritis 11-15 months before survey distribution

Exclusion Criteria:

* Legally incompetent citizens, i.e., persons with a legal guardian, will not be asked to participate.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be identified based on the NOMESCO (Nordic Medico-Statistical Committee) Classification of Surgical Procedures from the the Danish National Patient Register by using SKS-code the codes for THA patients will be SKS-code DM16 [hip osteoarthritis] + KNFB20 or KNFB30 or KNFB40[Primary Total Hip Arthroplasty]. For total knee arthroplasty (TKA), SKS-code DM17 [knee osteoarthritis] + KNGB20, KNGB30 or KNGB40 [primary total knee arthroplasty]. For medial unicompartmental knee arthroplasty (UKA), SKS-code DM17 [knee osteoarthritis] + KNGB01 or KNGB11 [primary medial unicompartmental knee arthroplasty].
Sampling Method: Non-Probability Sample
Enrollment: 6400 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Moderate/Severe Persistent Postoperative Pain | 11-15 months postsurgically
  The primary outcome is the number of patients with moderate or severe persistent postsurgical pain in the operated hip or knee, defined as patients with a numerical rating scale (NRS) score higher than 3.
  The outcome will be presented as Odd Ratio (OR) with its' corresponding 95% Confidence Interval (CI)

SECONDARY OUTCOMES:
Satisfaction | 11-15 months postsurgically
  Answering with "satisfied" or "very satisfied" in satisfaction question The outcome will be presented as Odd Ratio (OR) with its' corresponding 95% Confidence Interval (CI)
Willingness to repeat the surgery | 11-15 months postsurgically
  Answering "yes" in willlingness question The outcome will be presented as Odd Ratio (OR) with its' corresponding 95% Confidence Interval (CI)
Frequent pain | 11-15 months postsurgically
  Experiencing pain constantly, daily or few times a week The outcome will be presented as Odd Ratio (OR) with its' corresponding 95% Confidence Interval (CI)
Use of analgaesic | 11-15 months postsurgically
  The outcome will be presented as Odd Ratio (OR) with its' corresponding 95% Confidence Interval (CI)
Interference with daily activities | 11-15 months postsurgically
  Answering "some", "much" and "very much" in the interference question The outcome will be presented as Odd Ratio (OR) with its' corresponding 95% Confidence Interval (CI)
WOMAC pain score | 11-15 months postsurgically
  mean (standard deviaiton [SD]). We will report the mean difference (MD) and the corresponding 95% CI

CONTACTS AND LOCATIONS:
Overall Officials: Søren Overgaard, MD,DMSc,Prof, Study Director — Department of orthopedic surgery, Bispebjerg University Hospital, Denmark

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT06024161/Prot_SAP_000.pdf